CLINICAL TRIAL: NCT02669030
Title: A Six Week, Randomized, Double-Blind Placebo-Controlled, Suvorexant Augmentation Study of Antidepressant Treatment of Major Depressive Disorder With Residual Insomnia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Advanced Medical Research, Alpharetta, GA (Other)
Collaborators: Augusta University, Dept. of Psychiatry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVX-IIT2016-001
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Depression; Major Depressive Disorder; MDD; Insomnia
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suvorexant (Experimental): suvorexant 10mg/day, 15mg/day or 20mg/day augmentation of FDA-approved antidepressant treatment
  Interventions: Drug: suvorexant
- Placebo (Placebo Comparator): no augmentation of FDA-approved antidepressant treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: suvorexant — an FDA-approved sleep aid
  Other Names: Belsomra®
  Arms: Suvorexant
Drug: Placebo — control group
  Arms: Placebo

SUMMARY:
Depression with ongoing insomnia is a common clinical presentation with patients. Clinical data suggests that patients with insomnia that receive concomitant treatment with a sleep aid experience a more robust antidepressant response along with a quicker response. The purpose of this clinical study is to compare the effectiveness of the FDA-approved insomnia medication suvorexant, also known as Belsomra®, as add-on treatment to an antidepressant to that of placebo plus antidepressant treatment in patients with depression and residual or ongoing insomnia.

DETAILED DESCRIPTION:
Many patients with depression suffer from residual insomnia. This study is a six week, randomized, double-blind, placebo-controlled, trial to study suvorexant augmentation of continuing antidepressant therapy against placebo with continuing antidepressant therapy. Patient volunteers must be on a stable antidepressant treatment and will remain on this treatment for the duration of the study. Patient volunteers that qualify and enroll in the clinical trial will either receive suvorexant 10 mg/day and may have it adjusted to a dose of either 15 mg or 20 mg/day. Treatment is for a total of six weeks in addition to a clinical follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Provide written Informed Consent
* Diagnosis of depression (MDD)
* Currently on antidepressant
* Healthy and/or stable medically

Exclusion Criteria:

* unwilling to discontinue current use of sedative hypnotics/sleep aids/benzodiazepines or over the counter sleep aids/supplements
* currently using other psychotropics other than antidepressants
* at risk of self harm or a suicide attempt within the past 12 months
* history or presence of psychotic disorders
* known hypersensitivity to suvorexant
* presence of any other sleep disorder other than residual insomnia of depression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time | Six weeks ( baseline to end of treatment)
  assessment of total amount of time spent sleeping

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Six weeks ( baseline to end of treatment)
  assessment of insomnia severity
Hamilton Depression Rating Scale | Six weeks ( baseline to end of treatment)
  assessment fo depressive symptom severity
Sheehan Disability Scale | Six weeks ( baseline to end of treatment)
  assessment of impact of symptoms on performance
Wake After Sleep Onset (WASO) | Six weeks ( baseline to end of treatment)
  assessment of amount of time spent awake after initial onset of sleep
Sleep Latency (SL) | Six weeks ( baseline to end of treatment)
  assessment of amount of time it takes to fall asleep
Perceived Deficits Questionnaire (PDQ) | Six weeks ( baseline to end of treatment)
  a brief patient-rated scale to assess subjective cognitive dysfunction in people with depression

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Sambunaris, MD, Principal Investigator — Institute for Advanced Medical Research
Locations (2):
- United States (2):
  - Institute for Advanced Medical Research @ Mercer Univeristy, Atlanta, Georgia
  - Medical College of GA at Augusta Univeristy, Augusta, Georgia